CLINICAL TRIAL: NCT00946413
Title: Application and Evaluation of Group Cognitive Intervention for Depressed Adolescents
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: Department of Health (Ambiguous)
Responsible Party: Hsiu-Ju Chang, Taipei Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DOH95-TD-M-113-058
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Community Adolescents at Risk for Depression and Suicide
Keywords: CBT, Depressed and suicidal adolescents
MeSH Terms: conditions — Suicide; Color Vision Defects; Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT plus parent education (Experimental)
  Interventions: Behavioral: CBT plus parent education
- CBT alone (Experimental)
  Interventions: Behavioral: CBT alone

INTERVENTIONS:
Behavioral: CBT plus parent education — The 10-session group CBT with two-session parental education in our study was derived from the CWDA, with some modifications made based on cultural considerations. Skills taught and discussed included mood monitoring, improving social skills, increasing pleasant activities, decreasing anxiety, reducing depressogenic cognitions, improving communication, and conflict resolution. The issues taught and discussed included an introduction to adolescent depression and suicide, their etiology, symptoms, treatment, and prognosis, as well as stress management. A 1-year individual follow-up program was used to maintain the effect of the experimental intervention and to provide necessary individual interventions for students such as CBT, support, and counseling.
  Arms: CBT plus parent education
Behavioral: CBT alone — The 10-session group CBT with two-session parental education in our study was derived from the CWDA, with some modifications made based on cultural considerations. Skills taught and discussed included mood monitoring, improving social skills, increasing pleasant activities, decreasing anxiety, reducing depressogenic cognitions, improving communication, and conflict resolution.A 1-year individual follow-up program was used to maintain the effect of the experimental intervention and to provide necessary individual interventions for students such as CBT, support, and counseling.
  Arms: CBT alone

SUMMARY:
Cognitive behavioral therapy (CBT) is effective and CBT with parental involvement has potential in preventing and treating adolescent depression. The purpose of this study was to compare the short- and long-term effectiveness of CBT alone and CBT plus parental education for community-based adolescents at risk for depression and suicide in Taiwan. It is hypothesized that the CBT alone and CBT with parental education group are more effective than the control group.

DETAILED DESCRIPTION:
Cognitive behavioral therapy (CBT) is well known for its active, directive, time-limited, and structured approach. Despite an increasing prevalence of adolescent depression in Taiwan, few studies have been conducted to evaluate the immediate and long-term effectiveness of CBT for community-based adolescents at risk for depression and suicide. Also, little is known about the effectiveness of the involvement of parents in CBT groups. The Adolescent Coping with Depression Course (CWDA) (19) is an effective CBT-oriented group intervention for adolescent depression. However, it has not been tested in specific cultural groups. The primary purpose of this study was therefore to compare the immediate and long-term effectiveness of CBT alone, CBT with parental education, and control groups for community-based adolescents at risk for depression and suicide.A quasi-experimental research design was used in this study. Community-based high school students at risk for depression and suicide were recruited and assigned to one of two experimental groups or a control group. Students in the experimental groups received CBT plus parental education (group A, n = 9) or CBT alone (group B, n = 10). The control group was designed as a waiting list group (group C, n = 12). Both experimental groups received a follow-up session 1 year after the intervention. Several outcome variables (depressive symptoms, suicidal ideation, cognitive triad, learned resourcefulness [LR], and salivary cortisol level) were used to determine the effectiveness of treatment.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate group assignment and grant consents

Exclusion Criteria:

* unwilling to participate potential group activity and grant consents
* severe physical or psychiatric disorders

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
depressive symptoms, suicidal ideation, cognitive triad, learned resourcefulness (LR), and salivary cortisol | 6

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Ju Chang, phD, Principal Investigator — School of Nursing, Taipei Meidcal University
Locations (1):
- School of Nursing, Taipei Medical University, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://www.cachildwelfareclearinghouse.org/program/127/detailed#relevant-research